CLINICAL TRIAL: NCT06358924
Title: The Effect of Different Desensitizing Agents on Post-bleaching Hypersensitivity, Shade Stability and Surface Properties of Bleached Enamel. An In-vitro and In-vivo Study.
Brief Title: Effect of Different Desensitizing Agents on Post-bleaching Hypersensitivity and Shade Stability
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FDASU-RecID032004
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Tooth Hypersensitivity
Keywords: Dental Bleaching; Shade Stability
MeSH Terms: conditions — Dentin Sensitivity | interventions — potassium nitrate; Fluorides; Durapatite

STUDY DESIGN:
Intervention Model Description: This clinical study was conducted to evaluate the effect of using different desensitizing agents:
  1. As recommended by manufacturer
  2. Casein phosphopeptide-amorphous calcium phosphate/fluoride (CPP-ACPF) containing desensitizing agent
  3. Hydroxyapatite/fluoride/xylitol containing desensitizing agent
  4. Poly (amido amine) dendrimer with carboxylic acid terminal functional group containing desensitizing agent.
  On patients subjected to bleaching procedure using hydrogen peroxide containing bleaching agent.
  The clinical evaluation included:
  1. Post-bleaching hypersensitivity.
  2. Post-bleaching long-term shade stability.
Who Masked: Participant, Outcomes Assessor
Masking Description: This clinical trial was double blinded trial in which both the participant and outcome assessor were blinded to allocation, thus the participant was unaware of which experimental material had been assigned to him/her. Also the outcome assessors were blinded to the treatment that each participant had received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- After whitening mousse (Experimental): 30 % Xylitol, 4.2 % potassium nitrate, and 1450 ppm fluoride. Topical tooth gel Gel was applied on bleached teeth for 10 minutes according to manufacturer's instructions.
  Interventions: Other: Potassium nitrate with fluoride
- Mi Paste Plus (Experimental): Casein-phosphopeptide-amorphous calcium phosphate with 0.2 % sodium fluoride (900ppm) Topical tooth cream Cream was applied on bleached teeth for 3 minutes according to manufacturer's instructions
  Interventions: Other: Casein phosphopeptide-amorphous calcium phosphate with fluoride
- Hydroxyapatite and Fluoride (ReminPro) (Experimental): Hydroxyapatite (calcium and phosphate), ethanolic colophony, fluoride (1450 ppm NaF) and xylitol Topical water based tooth cream Cream was applied on bleached teeth for 3 minutes according to manufacturer's instructions
  Interventions: Other: Hydroxyapatite with fluoride
- PAMAM "poly (amido amine)" dendrimer (Experimental): PAMAM-succinamic acid dendrimer, 1,4-diaminobutane core, generation 4 solution. 10 wt.% in water Colorless liquid The liquid was applied on bleached teeth for 30 minutes (according to previous studies)
  Interventions: Other: PAMAM-carboxylic acid dendrimer

INTERVENTIONS:
Other: Potassium nitrate with fluoride — Bleaching of teeth using in-Office chemically-activated bleaching agent (Power Whitening YF) was performed followed by the application of the desensitizing agent recommended by the manufacturer (After Whitening Mousse), once for 10 minutes.
  Arms: After whitening mousse
Other: Casein phosphopeptide-amorphous calcium phosphate with fluoride — Bleaching of teeth using in-Office chemically-activated bleaching agent (Power Whitening YF) was performed followed by the application of Mi Paste Plus once for 3 minutes.
  Arms: Mi Paste Plus
Other: Hydroxyapatite with fluoride — Bleaching of teeth using in-Office chemically-activated bleaching agent (Power Whitening YF) was performed followed by the application of Hydroxyapatite and Fluoride (ReminPro) once for 3 minutes.
  Arms: Hydroxyapatite and Fluoride (ReminPro)
Other: PAMAM-carboxylic acid dendrimer — Bleaching of teeth using in-Office chemically-activated bleaching agent (Power Whitening YF) was performed followed by the application of PAMAM once for 30 minutes.
  Arms: PAMAM "poly (amido amine)" dendrimer

SUMMARY:
This study compared the effect of four different desensitizing agents on shade stability and dental hypersensitivity following dental bleaching procedure. The follow-up periods ranged from 24 hours to 1 year.

DETAILED DESCRIPTION:
This study was conducted to assess the effectiveness of 4 different desensitizing agents used after dental bleaching regarding dental hypersensitivity and shade stability. It was a double-blinded randomized clinical trial.

The ethical approval was obtained in May 2020 by the Research Ethics Committee an Institutional Review Board, Faculty of Dentistry, Ain Shams University (FDASU-REC).

The number of patients was determined according to G-Power program with a power (1-β error) of 0.8 (Power = 80%), and 95% confidence level (α = 0.05) using a two-sided hypothesis test. According to sample size calculation, 40 patients were needed for this study (n=10 per group).

Patients were selected according to inclusion and exclusion criteria and were randomly assigned into 4 groups according to the desensitizing agent used. The 4 desensitizing agents were: After Whitening Mousse, Mi Paste Plus, Hydroxyapatite and Fluoride (ReminPro) and PAMAM.

Patients signed an informed consent and received a detailed explanation of the study procedures. Baseline dental shade was recorded using Vita Easy-Shade spectrophotometer and Vita Classical Shade guide. Baseline sensitivity was assessed and recorded using a VAS.

All patients received dental bleaching using In-office chemically activated Power Whitening YF (WHITEsmile, Germany) followed by a desensitizing procedure using the desensitizing agent assigned to the specific experimental group.

Dental shade and dental hypersensitivity was assessed at different follow-up appointments; 24-hours, 3 days, 1 week, 1 month, 3 months, 6 months, 9 months and 1 year following the procedures.

Assessment of these variables at follow-up appointments was performed by 2 external assessors, and patients were blinded to the type desensitizing agent used.

ELIGIBILITY:
Inclusion Criteria:

* Participants with their entire upper and lower teeth, from right first premolar to left first premolar, present and sound, without restorations or periodontal disease.
* The participants had low-caries index scores.
* Participants had teeth with a Vita-color shade of A2 or darker.
* Cooperative behavior patient and medically free.
* Patient ages between 18 to 40 years old

Exclusion Criteria:

* Serious medically compromised patients.
* Smoking, alcoholism.
* Hypersensitivity to the agents used in the study.
* Lactating, pregnant patients.
* Patients with serious oral diseases, as acute necrotizing gingivitis, acute gingiva stomatitis, or those undergoing orthodontic treatment.
* Patients with dental enamel cracks.
* Patients who've had previous bleaching treatments

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2021-11-13 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Post-bleaching hypersensitivity | 24 hours, 3 days, 7 days, 1 month, 3 months, 6 months, 9 months and one year post bleaching
  Assessment was carried out by a visual analogue scale (VAS), from 0 (no tooth sensitivity at all) to 10 (intolerable pain). The air stimulus was applied at a distance of 0.5-1 cm for 2 seconds by the maximum power of the compressed air jet from the dental unit. Then patients were asked to describe the intensity of pain by numbers from 1 to 10.
  Sensitivity was measured before bleaching (baseline) and at each follow up period, 24 hours, 3 days, 7 days, 1 month, 3 months, 6 months, 9 months and one year post bleaching.
Shade stability | 24 hours, 3 days, 7 days, 1 month, 3 months, 6 months, 9 months and one year post bleaching
  Assessment was carried out using Vita Easy-Shade V. Two measurements were taken for each tooth from the upper right canine to the upper left canine, and same for the lower arch. For light condition standardization, all shade measurements were carried out under natural daylight in combination with constant artificial light sources; the clinic overhead lights in combination with the dental unit light directed away from the patient. The shade of each tooth was recorded as well as the values of L, a, and b. The shade of the upper two centrals was confirmed using Vita classical shade guide.
  Shade assessment was carried out before bleaching, and at each follow up period, 24 hours, 3 days, 7 days, 1 month, 3 months, 6 months, 9 months and one year post bleaching.

CONTACTS AND LOCATIONS:
Overall Officials: Farid MS El-Askary, Professor, Study Director — Faculty of Dentistry, Ain Shams University
Locations (1):
- Faculty of Dentistry, Ain Shams University, Cairo, El Weilli, Egypt

IPD SHARING:
Plan to Share IPD: No